CLINICAL TRIAL: NCT04032145
Title: Characterization of Health Conditions of Visitors of the Montreal Museum of Fine Arts: A Prevalence Survey
Brief Title: Characterization of Health Conditions of Visitors of the Montreal Museum of Fine Arts
Status: Completed | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: 2020-1878
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Prevention; Health Promotion
Keywords: Prevention, museum, art

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: All participants who go to the Montreal Museum of Fine Arts will fill out an online questionnaire called: CESAM ( Self Administered Questionnaire). This questionnaire will asse participant's health condition. Moreover, the goal of the questionnaire is to evaluate if art activities may change the participants' health conditions in time.

SUMMARY:
This study evaluates the effects of arts on the Montreal Museum's clients.

DETAILED DESCRIPTION:
Acting early in the process of weakening elders in order to keep them longer in good health and socially active is possible. During the past decade, museums have become involved in the care of patients by using art to improve their quality of life and well-being. Museums have, thus, emerged as new partners in public health. Very few programs developed by museums have focused on elders. Only one focused on elders in situation of early frailty and demonstrated that it was possible, through participatory visual art-based activities, to improve the health status of elders living at home.

ELIGIBILITY:
Inclusion Criteria:

* Being 50 years old
* Coming at Montreal Museum of Fine Arts for guided visits, arts activities, and so forth.

Exclusion Criteria

-No internet connection and electronic device like cell phone, Ipad or computer.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Montreal Museum's clients will be invited to participate in this study, and if they accept to be a part of it, we will ask them to fill out an online questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Health Condition | one month
  Health condition will be evaluates based on a questionnaire called: CESAM(Self Administered Questionnaire). This is an assessment questionnaire that each participant will answer once. The questionnaire is designed that participant's answers to questions are scored. After the answers are summed , the Principal Investigator will obtain an overall measure of participant' health condition.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada